CLINICAL TRIAL: NCT00234104
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Dose Response of OPC-41061 in Congestive Heart Failure Patients With Extracellular Volume Expansion
Brief Title: A Dose-finding Study of OPC-41061 in Treatment of Cardiac Edema (Congestive Heart Failure)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-03-001; JapicCTI-050038
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Heart Failure, Congestive; Edema
Keywords: OPC-41061; Tolvaptan; Heart Failure; Edema; Extracellular volume expansion
MeSH Terms: conditions — Heart Failure; Edema | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: OPC-41061(Tolvaptan)

SUMMARY:
This drug is being developed to treat cardiac edema. The primary purpose of this study is to investigate the dose response for body weight in seven-day repeated oral administration of OPC-41061 at 15, 30, and 45 mg or placebo in patients with extracellular volume expansion secondary to CHF despite taking furosemide at 40 mg/d or more. This study is being conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CHF who exhibit edema, jugular venous distention, hepatomegaly, pulmonary congestion, or 3rd sound due to extracellular volume expansion
2. Hospitalized patients or patients who can be hospitalized for the study from the commencement of the observation period to the end-of-study examination
3. Men and women between the ages of 20 and 80 (non-inclusive) at the time of giving consent
4. Patients who have taken furosemide at 40 mg/d or more (oral dosing) without alteration of dosage for the 3 days of the observation period
5. Patients whose body weight has been stable (±1.0 kg) for 2 days prior to commencement of study drug administration

Exclusion Criteria:

1. Patients with unstable heart failure (acute heart failure, acute exacerbation of chronic heart failure, etc)
2. Patients with an implanted ventricular assist device
3. Patients who have undergone or are scheduled to undergo any of the following procedures

   * Heart surgery involving thoracotomy within 60 days prior to the screening examination
   * Pacemaker implant surgery involving bilateral pacing within 60 days prior to the screening examination
   * Angioplasty, electrophysiologic device implantation, ventricular assist device implantation, heart transplant, or other cardiac surgery scheduled within 30 days after the screening examination
4. Patients with any of the following diseases, complications, or symptoms

   * Suspected hypovolemia
   * Onset of acute myocardial infarction within 30 days prior to the screening examination
   * Hypertrophic cardiomyopathy (excluding diastolic phase)
   * Definitively diagnosed active myocarditis or amyloid cardiomyopathy
   * Valvular heart disease with significant stenosis
   * Untreated thyroid disease
   * Progressive neurological disease (Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc) or severe episodic neurological disease (epilepsy, Guillain-Barre syndrome, etc)
   * Diabetes with poor glycemic control
   * Anuria
   * Hepatic coma
   * Hyponatremia of moderate or greater severity (serum Na < 120 mEq/L)
5. Patients with a history of the following conditions

   * Occurrence of sustained ventricular tachycardia or ventricular fibrillation within 30 days prior to the screening examination (except for patients using an implantable cardioverter-defibrillator)
   * Evident cerebral infarction
   * Multiple stroke
   * Occurrence of a cerebrovascular accident within 30 days prior to the screening examination
   * Hypersensitivity or idiosyncratic reaction to benzazepine derivatives, such as benazapril
6. Patients with a history of drug abuse or alcoholism in the past year
7. Patients in a state of morbid obesity with a body mass index (weight[kg] ÷ height [m]2) over 35
8. Patients with a supine systolic arterial blood pressure of less than 90 mmHg
9. Patients with any of the following abnormal laboratory values: Hemoglobin <9 g/dL, total bilirubin >3.0 mg/dL, serum creatine >3.0 mg/dL, serum Na >147 mEq/L, or serum K >5.5 mEq/L
10. Patients not capable of taking oral medication
11. Patients who are nursing, pregnant, capable of pregnancy, or intending to become pregnant during or shortly after the study period
12. Patients who have taken a study drug other than OPC-41061 within 30 days prior to screening
13. Patients who have previously taken OPC-41061 in this study or another study of OPC-41061
14. Patients otherwise judged by the principal investigator or attending investigator to be inappropriate for inclusion in the study (eg, patients with hepatic cirrhosis, renal disease, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: OPC-41061 0 mg/day
- 15 mg of OPC-41061: OPC-41061 15 mg/day
- 30 mg of OPC-41061: OPC-41061 30 mg/day
- 45 mg of OPC-41061: OPC-41061 45 mg/day
Period: Overall Study
Arm/Group | Placebo | 15 mg of OPC-41061 | 30 mg of OPC-41061 | 45 mg of OPC-41061
Started | 30 | 29 | 34 | 29
Completed | 26 | 28 | 29 | 21
Not Completed | 4 | 1 | 5 | 8
Not completed — Adverse Event | 4 | 0 | 3 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: 1 Subject of each arm were excluded form the analysis set because emergency codes were lost.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 15 mg of OPC-41061 | 30 mg of OPC-41061 | 45 mg of OPC-41061 | Total
Number analyzed (Participants) | 29 | 28 | 33 | 28 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 11 | 14 | 46
  >=65 years | 18 | 18 | 22 | 14 | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.4) | 66.9 (9.6) | 66.4 (12.5) | 62.6 (12.5) | 66.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 8 | 4 | 36
  Male | 18 | 15 | 25 | 24 | 82
Region of Enrollment [Number; unit: participants]
  Japan | 29 | 28 | 33 | 28 | 118

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: The body weight change from baseline following final trial drug administration
Time Frame: Baseline, at the time of final trial drug administration
Population: 1 Subject of Placebo arm who experienced a serious adverse event was excluded from efficacy analysis set because the emergency code was broken.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | 15 mg of OPC-41061 | 30 mg of OPC-41061 | 45 mg of OPC-41061
Number analyzed (Participants) | 28 | 28 | 33 | 28
Kg | -0.53 (0.96) | -1.62 (1.55) | -1.35 (1.54) | -1.85 (1.10)
Statistical Analysis 1: Comparison: Placebo vs 15 mg of OPC-41061; Test type: Superiority or Other; p = 0.0074, t-test, 2 sided; Dunnett's test was used; Mean Difference (Final Values) = -1.09
Statistical Analysis 2: Comparison: Placebo vs 30 mg of OPC-41061; Test type: Superiority or Other; p = 0.0459, t-test, 2 sided; Dunnett's test was used; Mean Difference (Final Values) = -0.82
Statistical Analysis 3: Comparison: Placebo vs 45 mg of OPC-41061; Test type: Superiority or Other; p = 0.0010, t-test, 2 sided; Dunnett's test was used; Mean Difference (Final Values) = -1.32

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Placebo | 15 mg of OPC-41061 | 30 mg of OPC-41061 | 45 mg of OPC-41061
Serious Adverse Events (participants affected / at risk) | 4/29 | 0/28 | 1/33 | 2/28
Other Adverse Events (participants affected / at risk) | 14/29 | 21/28 | 25/33 | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | 15 mg of OPC-41061 (N=28) | 30 mg of OPC-41061 (N=33) | 45 mg of OPC-41061 (N=28)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | 15 mg of OPC-41061 (N=28) | 30 mg of OPC-41061 (N=33) | 45 mg of OPC-41061 (N=28)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Thirst (General disorders) | 3 (3) | 6 (6) | 9 (9) | 15 (15)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood Osmolarity Increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Blood Potassium Increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Blood Pressure Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood Pressure Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Urea Increased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Blood Uric Acid Increased (Investigations) | 0 (0) | 6 (7) | 4 (4) | 2 (2)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Protein Urine Present (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 6 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No